CLINICAL TRIAL: NCT00374140
Title: Phase II Trial of RAD001 (Everolimus) in Previously Treated Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ahmad Tarhini (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Ahmad Tarhini, Study Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-049
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell; lung
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Everolimus) (Experimental): RAD001 (Everolimus)10 mg by mouth daily without interruption
  Interventions: Drug: RAD001 (everolimus)

INTERVENTIONS:
Drug: RAD001 (everolimus) — 10 mg by mouth daily without interruption for 3-week cycles until disease progression or intolerable toxicities
  Other Names: Certican®

SUMMARY:
This is a phase II, two-stage, open-label, single-agent study of the experimental drug RAD001 (everolimus) in patients with previously treated small cell lung cancer. RAD001 will be administered orally at a dose of 10 mg daily.

DETAILED DESCRIPTION:
This is a phase II, two-stage, open-label, single-agent study of the experimental drug RAD001 (everolimus) in patients with previously treated small cell lung cancer. Patients may have received up to 2 prior chemotherapy regimens for small cell lung carcinoma, but no prior therapy with an m-TOR inhibitor. RAD001 will be administered orally at a dose of 10 mg daily. A cycle will be defined as 3 weeks of study drug administration, and patients will have tumor measurements every 2 cycles. Study participation will continue until disease progression or intolerable toxicities. In addition, in patients who consent, archival tumor tissue (paraffin block from original biopsy) will be collected for research purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed small cell carcinoma of the lung that has progressed post first-line therapy. Mixed small and non-small cell tumors are excluded.
2. Prior chemotherapy for small cell carcinoma. Up to 2 prior chemotherapy regimens for small cell lung carcinoma are allowed. No prior therapy with an m-TOR inhibitor (e.g. CCI-779).
3. Unidimensionally measurable disease (RECIST criteria). If the only site of measurable disease is in a previously irradiated area, the patient must have documented progression of disease in this area.
4. ECOG performance status 0-2.
5. A minimum of 4 weeks should elapse from prior chemotherapy. Patients must have fully recovered from the effects of any prior surgery or radiation therapy or other anticancer therapies, including immunotherapy and investigational agents.
6. No progressive brain metastases. Brain metastases should have been previously treated with surgery and/or radiation.
7. Patients with a prior malignancy should have at least 3 years of disease-free survival. Prior curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer or other in situ malignancies are allowed.
8. No other coexisting medical condition that would preclude full compliance with the study.
9. Required laboratory values (obtained < 1 week prior to enrollment):

   * ANC >/= 1500/mm³
   * Platelets >/= 100,000/mm³
   * AST and ALT ≤ 3 x ULN (upper limits of normal). In patients with liver metastases AST and ALT should be < 5 x ULN.
   * Total bilirubin up to 1.5 x ULN (upper limits of normal).
10. Age >/= 18 years and capacity to give informed consent.
11. Patients should be advised to discontinue drugs that interact with CYP3A4 (see list of examples in Table 3.1 of the full protocol), if medically safe.
12. All patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

1. Prior treatment with any investigational agent within the preceding 4 weeks.
2. Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmias active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper GI tract ulceration).
3. A known history of HIV seropositivity.
4. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
5. Patients with an active, bleeding diathesis or on anticoagulation (except low dose warfarin).
6. Pregnant and lactating women are excluded from the study because the agents used in this study may be teratogenic to a fetus and there is no information on the excretion of the agents or their metabolites into breast milk.
7. Women of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study.
8. Patients should not be on chronic systemic glucocorticoids or other immunosuppressant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (19):
- United States (19):
  - UPMC Cancer Center - Teramana Cancer Center - Steubenville, Steubenville, Ohio
  - UPMC Cancer Center - Beaver, Beaver, Pennsylvania
  - UPMC Cancer Center - Clairton, Clairton, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion - Greensburg, Greensburg, Pennsylvania
  - UPMC Cancer Center - Oakbrook Commons - Greensburg, Greensburg, Pennsylvania
  - UPMC Cancer Center - Indiana, Indiana, Pennsylvania
  - UPMC Cancer Center - John P. Murtha Pavilion - Johnstown, Johnstown, Pennsylvania
  - UPMC Cancer Center - McKeesport, McKeesport, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Cancer Center - Sewickley Medical Oncology/Hematology Group, Moon Township, Pennsylvania
  - UPMC Cancer Center - New Castle, New Castle, Pennsylvania
  - UPMC Cancer Center - St. Margaret's, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Mercy, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Passavant, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Upper St. Clair, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center - Washington, Washington, Pennsylvania
  - UPMC Cancer Center - North Hills, Wexford, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RAD001 (Everolimus)
Started | 40
Completed | 38
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | RAD001 (Everolimus)
Number analyzed (Participants) | 40
Age, Customized [Median (Full Range); unit: years] | 64 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Determine the Proportion of Previously Treated Small Cell Lung Cancer (SCLC) Patients Whose Disease Has Not Progressed Following 6-weeks (2 Cycles) of Treatment With RAD001.
Time Frame: Two cycles of treatment with RAD001 (~6 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001 (Everolimus)
Number analyzed (Participants) | 35
percentage of participants | 26 [11 to 40]

2. Secondary Outcome: Overall Survival
Time Frame: From entry in trial to up to 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 (Everolimus)
Number analyzed (Participants) | 40
months | 6.7 [4.0 to 8.6]

3. Secondary Outcome: Progression-free Survival
Time Frame: From entry into trial to up to 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 (Everolimus)
Number analyzed (Participants) | 35
months | 1.3 [1.3 to 1.4]

4. Secondary Outcome: Objective Response Rate
Description: Number of patients for which response to treatment was observed / total number of patients.
Time Frame: From beginning of treatment up to 60 months
Population: Evaluable for response included patient had completed at least one cycle of therapy with everolimus.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001 (Everolimus)
Number analyzed (Participants) | 35
percentage of participants | 3 [0 to 8]

ADVERSE EVENTS:
Arm/Group | RAD001 (Everolimus)
Serious Adverse Events (participants affected / at risk) | 18/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (Everolimus) (N=40)
Death due to progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4
Confusion (Psychiatric disorders) | 2
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5
Gastrointestinal Fistula (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Infection with normal ANC or grade 1 or 2 Neutrophils (Infections and infestations) | 3
Somnolence (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (Everolimus) (N=40)
Constitutional (General disorders) | 12
Gastrointestinal (Gastrointestinal disorders) | 20
Increased transaminases (Hepatobiliary disorders) | 3
Infection (without neutropenia) (Infections and infestations) | 5
Metabolic (Metabolism and nutrition disorders) | 7
Lethargy, confusion (Nervous system disorders) | 2
Dyspnea, pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Increased creatinine (dehydration) (Renal and urinary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Anemia (Blood and lymphatic system disorders) | 9
Neutropenia (Investigations) | 13
Thrombocytopenia (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes